CLINICAL TRIAL: NCT05358483
Title: The PROMISE Study: PROspective Study of Mothers' and Infants' Social and Epidemiologic Determinants of Health
Brief Title: PROspective Study of Mothers' and Infants' Social and Epidemiologic Determinants of Health
Acronym: PROMISE
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Jungheim, Chief of Reproductive Endocrinology and Infertility in the Department of Obstetrics and Gynecology, Northwestern University
Other Study IDs: STU00215252
Record Dates: First submitted 2021-12-15; First posted 2022-05-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the PROMISE study is to determine how pre-conception lifestyle factors (e.g., sleep, nutrition, physical activity) affect short- and long-term reproductive outcomes.

DETAILED DESCRIPTION:
The overall goal of the PROMISE study is to identify strategies to improve health outcomes for women and their children. The proposed study is important and novel as it aims to capture women before they are pregnant. Current research on maternal and child health often focuses on women who are already pregnant. This time period is likely too late to make a meaningful clinical impact on long term maternal and child health outcomes influenced by social and epidemiologic determinants of health as important epigenetic changes are or have already taken place. Examples of tools that will be used to capture social and epidemiologic data include validated surveys for nutrition, physical activity, sleep, and stress. The importance of these tools is that many of the data points captured are modifiable, and therefore if associations are noted between these data points and health outcomes, actionable interventions may be developed and implemented for women who are preconceptional.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-44 seeking pregnancy at Northwestern Fertility and Reproductive Medicine (FRM) who agree to

  1. Be followed for a period for up to 25 years
  2. Share information regarding their child's health
* No prior IVF cycles

Exclusion Criteria:

* Women using donor oocytes or gestational carriers
* Inability or unwillingness to provide informed consent for any aspects of the study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The PROMISE Study is enrolling women undergoing IVF for the first time without use of a gestational carrier or donor oocytes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2046-12 (Estimated); Study Completion 2046-12 (Estimated)

PRIMARY OUTCOMES:
Live birth after embryo transfer | ~0-24 months
  Live birth after embryo transfer (y/n)

SECONDARY OUTCOMES:
Cycle number | ~0-24 months
  IVF cycle number
AMH | ~0-24 months
  Most recent AMH
Antral follicle count (AFC) | ~0-24 months
  Most recent AFC
Diagnosis/reason for ART | ~0-24 months
  E.g., male factor, DOR, tubal factor
Stimulation type | ~0-24 months
  Antagonist, microcode flare, long agonist, minimal stimulation
Total gonadotropin dose (IU/L) | ~0-24 months
  Total gonadotropin dose
Maximum estradiol level (pmol/L) | ~0-24 months
  Maximum estradiol level
Days of stimulation | ~0-24 months
  Total number of days of stimulation
Trigger type | ~0-24 months
Sperm source | ~0-24 months
Number follicles >14 mm | ~0-24 months
Cycle cancellation | ~0-24 months
  Cycle cancellation (Y/N). If Y, reason for cancellation
Number of oocytes retrieved | ~0-24 months
Number of mature oocytes | ~0-24 months
Number of blastocysts | ~0-24 months
Number of embryos transferred | ~0-24 months
Day of embryo transfer | ~0-24 months
Type of embryo transfer | ~0-24 months
  Frozen or fresh embryo transfer
Frozen embryo transfer protocol | ~0-24 months
Luteal phase support | ~0-24 months
Number of embryos cryopreserved | ~0-24 months
Stage of embryo cryopreservation | ~0-24 months
Grade of embryo transferred | ~0-24 months
PGT | ~0-24 months
PGT indication | ~0-24 months
PGT methodology | ~0-24 months
Endometrial thickness | ~0-24 months
Ovarian hyperstimulation syndrome | ~0-24 months
Clinical outcome | ~0-24 months
Insemination Type | ~0-24 months
  ICSI, conventional, split
Singleton pregnancy | ~12-36 months
Multiple gestation | ~12-36 months
Asthma | ~12-36 months
Gestational diabetes | ~12-36 months
Insulin | ~12-36 months
Gestational hypertension/pre-eclampsia | ~12-36 months
Abruption | ~12-36 months
Placental disorders | ~12-36 months
  Placenta accreta, Placenta previa, Placenta increta, Placenta percreta
Intrauterine growth restriction | ~12-36 months
Congenital malformation | ~12-36 months
  Cleft palate, genetic defect, limb defect, cardiac defect, other
Thyroid disease | ~12-36 months
Heart disease | ~12-36 months
Renal disease | ~12-36 months
Polyhydramnios | ~12-36 months
Lupus | ~12-36 months
Clinical chorioamnionitis | ~12-36 months
Prenatal genetic testing | ~12-36 months
Type of prenatal genetic testing | ~12-36 months
  NIPT, CVS, amniocentesis
Maternal blood type | ~12-36 months
Preconception COVID vaccination | ~12-36 months
Pregnancy COVID vaccination | ~12-36 months
Predelivery hospitalization | ~12-36 months
Maternal weight at oocyte retrieval | ~12-36 months
  Weight (lbs)
Maternal height at oocyte retrieval | ~12-36 months
  Height (inches)
Number of mature oocytes inseminated | ~0-24 months
Number of mature oocytes fertilized (2PN) | ~0-24 months
Maternal weight at embryo transfer | ~12-36 months
Maternal weight at last OB visit | ~12-36 months
Maternal weight at 1 year postpartum | ~12-36 months
Date of delivery | ~12-36 months
Time of delivery | ~12-36 months
Weight at delivery | ~12-36 months
Mode of delivery | ~12-36 months
Preterm birth | ~12-36 months
  Birth <37 weeks
Spontaneous preterm birth | ~12-36 months
Presentation of spontaneous preterm birth (if applicable) | ~12-36 months
Tocolytic medication during pregnancy | ~12-36 months
Gestational age at delivery | ~12-36 months
Presentation of term birth (if applicable) | ~12-36 months
Magnesium sulfate administered | ~12-36 months
Intrapartum antibiotics | ~12-36 months
Length of hospital stay | ~12-36 months
Head circumference | ~12-36 months
Maternal mortality | ~12-36 months
Infection | ~12-36 months
Anesthetic complication | ~12-36 months
Antepartum hemorrhage | ~12-36 months
Postpartum hemorrhage | ~12-36 months
Blood transfusion | ~12-36 months
Thromboembolism | ~12-36 months
Birthweight | ~12-36 months
Small-for-gestational age | ~12-36 months
Large-for-gestational age | ~12-36 months
1-min APGAR score | ~12-36 months
5-min APGAR score | ~12-36 months
Arterial umbilical cord pH | ~12-36 months
Breastfeeding compliance | ~12-48 months
Postpartum weight change | ~12-48 months
General well-being | ~12-48 months
Length of NICU stay | ~12-48 months
Neonatal death | ~12-48 months
  <28 days post delivery
Breastfeeding | ~12-48 months
Supplemental formula | ~12-48 months
Breastfeeding at 1 year of life | ~12-48 months
Child weight at 1 year of life | ~12-48 months
Child height at 1 year of life | ~12-48 months
NICU admission | ~12-48 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily Jungheim, MD, MCSI, Principal Investigator — Division Chief of Reproductive Endocrinology and Infertility
Locations (1):
- Northwestern Medicine Fertility and Reproductive Medicine, Chicago, Illinois, United States